CLINICAL TRIAL: NCT01524419
Title: Women's Involvement In Decision Making At Labor And Its Effect on Their Perceived Labor Process
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0004-12-HYMC
Record Dates: First submitted 2012-01-25; First posted 2012-02-02 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-01

CONDITIONS: Mother (Person)
Keywords: spontaneous labor; term; surgical; mechanical; fetal or maternal complications

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women after vaginal birth

SUMMARY:
1. Increased women's involvement in decision making at labor process correlates with a positive perception of the labor process.
2. Increased maternal satisfaction with midwifery and gynecological care at labor correlates with a more positive perception of the labor process.

DETAILED DESCRIPTION:
The Interrelationship Between Women's Involvement In Decision Making In Labor And Their Perception Of The Labor Experience Labor is one of the most significant events in women's lives. The process and outcome of labor may have long term effects on the way women perceive the parenting role and their personal, emotional and physical capability. Each woman arrives to labor with a planned construct of beliefs, expectations and fantasies regarding the labor process and outcomes, which are driven from different cultural values and personal beliefs. The clinical reality does not always correlate with this emotional construct and with a woman's anticipated level of involvement in decision making at labor. Discrepancy between women's desired or expected labor processes and what happens in actuality may have a substantial impact on women's lives and on the way they will experience future births. The main goal of this research is to investigate the effects of labor process on women by examining the question whether women's involvement in decision making during labor has an effect on their perceived labor process.

The perceived labor process is a combination of a woman's level of engagement in decision making at labor, her perceived level of control in the labor process and the level of satisfaction from the obstetric caregivers (gynecologists and midwives). The participants of this research project shall be comprised of 100 women who were hospitalized during the two days immediately following labor and delivery in the maternity unit at Hillel Yaffe hospital, who gave birth in a normal delivery, at term (37 weeks of gestation) with no surgical or instrumental intervention and had no complications either to them or their babies. The participants will be given a self-replying questionnaire constructed especially for the purposes of this research project. The questionnaire is comprised of seven parts: (1) social-demographic information,(2) health background,(3) obstetric background,(4) the woman's perspective of labor process in general,(5) the woman's perspective of the progression of her actual labor,(6) the woman's evaluation of the attitude of obstetric caregivers (gynecologists and midwives) and (7) the level of control the woman had in decision making during labor and her perception of the labor experience. The research findings will be analyzed statistically using Statistical Package for the Social Sciences (SPSS) format. In addition to understanding the way women perceive their labor and delivery in terms of the level of involvement in decision making, these findings may also contribute to develop a therapeutic intervention tool to assist accommodating specific treatment to women in labor and childbirth according to the level of her desired involvement in decision making at birth, her viewpoint of therapeutic intervention and her expectations of the labor process.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal labor
* At term
* Hebrew/Arabic speakers

Exclusion Criteria:

* Mechanical or surgical intervention
* Maternal or fetal complications

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: women after vaginal birth at term with no mechanical or surgical intervention and with no maternal or fetal complications
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Merav Amos Chen, BA, Study Director — Hillel Yaffe Medical Center; Mordechai Hallak, prof, Principal Investigator — Hillel Yaffe Medical Center; Elad Mei-Dan, dr, Study Director — Hillel Yaffe Medical Center; Mally ehrenfeld, prof, Study Director — University of Tel-Aviv; Tammy Schifter, dr, Study Director — University of Tel-Aviv
Locations (1):
- Department of Obstetrics and Gynecology, Hillel-Yaffe Medical Center, Hadera, Israel, Israel